CLINICAL TRIAL: NCT05150665
Title: Evaluation of Mini and Macro-esthetics Following En- Masse Retraction Versus Two Step Retraction in Maxillary Protrusion Cases: A Randomized Clinical Trial
Brief Title: Evaluation of Mini and Macro-esthetics Following En- Masse Retraction Versus Two Step Retraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Sara Usama Saeed Imam, Principle Investigator, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUE.REC(26)/12-2019
Record Dates: First submitted 2021-11-26; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Bimaxillary Protrusion
Keywords: Mini-esthetics; Macro-esthetics; En-masse Retraction; Two step retraction; Extra-oral photographs; Adobe photoshop CC 2017 software; Lateral Cephalometric Radiographs

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Only the outcome assessors will be blind. The patients name will be sealed from pre and post photographs and cephalometric radiographs. Then two assessors will carry out, blindly and independently, the measurements and analysis of the study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- En-Masse Retraction (Experimental): Six anterior teeth (en-Masse) retracted using a crimpable hook distal to the upper lateral incisor and a power chain
  Interventions: Procedure: En-masse retraction
- two step retraction (Experimental): Six anterior teeth are retracted by two step technique by canine retraction followed by four anterior teeth retraction using a crimpable hook distal to the upper lateral incisor and a power chain
  Interventions: Procedure: Two step Retraction

INTERVENTIONS:
Procedure: En-masse retraction — Power chain and Crimpable hook for En-Masse Retraction Retraction will start on a 0.017"x0.025" Stainless steel wire using elastomeric chain (force applied will be 200 g per side) extending between the crimpable hooks and the miniscrew
  Arms: En-Masse Retraction
Procedure: Two step Retraction — Retraction of canine started on a 0.017"x0.025" Stainless steel wire using elastomeric chain (force applied will be 150 g per side)followed by anterior teeth retraction on 0.017"x0.025" Stainless steel wire using elastomeric chain (force applied will be 160 g per side) extending between the crimpable hooks and the mini-screw.
  Arms: two step retraction

SUMMARY:
There's a scarcity in literature concerning mini-esthetics specially maxillary gingival display changes following en-masse retraction and two-step retraction. The purpose of this study is to determine, In orthodontic patients with maxillary protrusion, which technique of retraction will result in better esthetics upon smiling following en-masse retraction or two step retraction mechanics.

DETAILED DESCRIPTION:
This study will be conducted in order to evaluate which technique of retraction will provide better outcome regarding mini and macro esthetics. In terms of mini esthetics, posed smiles will be analyzed to evaluate maxillary gingival display, as well as the analysis of smile arc, buccal corridor, inter-labial gap. In terms of macro esthetics, frontal and profile poses will be assessed to evaluate the nasolabial angle, mentolabial angle and upper and lower lip protrusion/ E- plane.

ELIGIBILITY:
Inclusion Criteria:

* Adults and Adolescent patients (both genders)
* Age range (16-24)
* Patients with maxillary protrusion requiring first premolars extraction (Bimaxillary Protrusion or Class II division 1 cases).
* Patients with fully erupted permanent teeth (not necessarily including the third molar).
* Cases requiring maximum anchorage during retraction.
* Good general and oral health

Exclusion Criteria:

* Patients suffering from any neural disorders or systemic diseases interfering with tooth movement.
* Patients with soft tissue problems such as cleft-palate patients
* Patients with extracted or missing permanent teeth. (except for third molars).
* Patients with badly decayed teeth.
* Patients with any parafunctional habits (i.e. Bruxism, tongue thrusting, mouth breathing, etc....).
* Patients with previous orthodontic treatment.

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2021-12-28 (Estimated); Study Completion 2021-12-28 (Estimated)

PRIMARY OUTCOMES:
Mini-esthetics including | From pre to post retraction (an average of 6 - 8 months)]
  Evaluation of (maxillary gingival display, Smile arc, buccal corridor) from social smile photograph Evaluation of (inter-labial gap) from At Rest photograph All primary outcome characteristics will be measured before and after retraction (measured Linear/ horizontal/ vertical in millimeters) by Adobe Photoshop CC 2017 software.

SECONDARY OUTCOMES:
Macro-esthetics evaluation of profile photograph including | upto 6 months from the start of orthodontic treatment.
  1. Nasolabial angle. 2. Mentolabial angle. 3. Incisors Inclination (Angular measurement in degrees). 4. Upper lip protrusion/ E- plane. 5. Lower lip protrusion/ E- plane. (Linear measurement in millimeters.) Cephalometric radiographs and Adobe Photoshop CC 2017 software

CONTACTS AND LOCATIONS:
Overall Officials: Yehya mostafa, Professor and chairman, Study Director — Future University in Egypt
Locations (1):
- Future University In Egypt, Cairo, Egypt